CLINICAL TRIAL: NCT00590408
Title: Efficacy and Safety of Coenzyme Q10 in the Treatment of Statin-Associated Myalgia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Creighton University (Other)
Responsible Party: Robyn Kondrack, PharmD, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-13642; 05-13642
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Statin-associated Myalgia
Keywords: coenzyme Q10; statin; myalgia
MeSH Terms: conditions — Myalgia | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: coenzyme Q10
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: matching placebo

INTERVENTIONS:
Dietary Supplement: coenzyme Q10 — 60mg capsule twice daily for 12 weeks
  Arms: 1
Dietary Supplement: matching placebo — matching placebo capsule twice daily for 12 weeks
  Arms: 2

SUMMARY:
Statins are medications that lower blood cholesterol by inhibiting cholesterol production in the liver. Overall, statins are well tolerated. Approximately 10% to 15% of patients report muscle aches/pain while taking statins. In a very small percentage of patients (<0.01%; less than one in 10,000 people), muscle aches/pains may be accompanied by more serious muscle damage. In these patients, statins must be discontinued. In some reports, patients taking statins have reduced blood levels of coenzyme Q10. Coenzyme Q10 is an essential protein which is present in all human cells needed for normal cell function. Coenzyme Q10 has been tested in patients with heart failure where it has been shown to be safe and effective. Many patients with heart conditions take coenzyme Q10, but the risks and benefits of supplementation with this product is unknown. Coenzyme Q10 is considered a dietary supplement and is not approved by the Food and Drug Administration (FDA) for any medical condition. Coenzyme Q10 has very few, if any, side effects. Upset stomach (gastritis), headache, body ache, and low blood pressure have been reported. The objectives of this project are to test the efficacy and safety of coenzyme Q10 in treating muscle aches/pain in patients already taking statins who develop these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are taking statins and develop unexplained, persistent myalgia with a normal plasma creatinine kinase level

Exclusion Criteria:

* Women of childbearing potential
* Patients currently taking coenzyme Q10 (or have taken in the previous 30 days)
* Patients receiving concomitant niacin, fibric acid derivatives, bile acid sequestrants, or other drugs that effect cholesterol levels or interact with statins
* Patients with a history of alcoholism or malnutrition
* Patients who have had acute coronary syndrome or muscle trauma in the prior 7 days
* Patients with a history of chronic muscle/joint pain, fibromyalgia, or degenerative disk disease.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy coenzyme Q10 in the treatment of myalgia in patients receiving statin therapy | every 3-5 days during the first week 2 weeks, then at 4 weeks and 12 weeks

SECONDARY OUTCOMES:
evaluate the safety of coenzyme Q10 in the treatment of myalgia in patients receiving statin therapy | every 3-5 days during the first week 2 weeks, then at 4 week and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Kondrack, PharmD, Principal Investigator — Creighton University
Locations (1):
- The Cardiac Center of Creighton University Medical Center, Omaha, Nebraska, United States